CLINICAL TRIAL: NCT00383448
Title: Treatment of High Risk, Inherited Lysosomal And Peroxisomal Disorders by Reduced Intensity Hematopoietic Stem Cell Transplantation
Brief Title: HSCT for High Risk Inherited Inborn Errors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2006-14; 0606M87246 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Adrenoleukodystrophy; Metachromatic Leukodystrophy; Globoid Cell Leukodystrophy; Tay Sachs Disease; Sandhoffs Disease; Wolman Disease; I-Cell Disease; Sanfilippo Syndrome; GM1 Gangliosidosis
Keywords: Stem cell transplantation; Inborn errors of metabolism; Adrenoleukodystrophy (ALD); Metachromatic leukodystrophy (MLD); Globoid cell leukodystrophy (GLD or Krabbe); Tay Sachs; Sandhoff; Sanfilippo syndrome; Mucopolysaccharidosis III (MPS-III); GM1 gangliosidosis; I-cell; mucolipidosis
MeSH Terms: conditions — Adrenoleukodystrophy; Leukodystrophy, Metachromatic; Leukodystrophy, Globoid Cell; Tay-Sachs Disease; Sandhoff Disease; Wolman Disease; Mucolipidoses; Mucopolysaccharidosis III; Gangliosidosis, GM1; Metabolism, Inborn Errors | interventions — Clofarabine; Whole-Body Irradiation; Melphalan; Hematopoietic Stem Cell Transplantation; Alemtuzumab; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated Patients (Experimental): Patients receiving chemotherapy (Hydroxyurea, Alemtuzumab, Clofarabine, Melphalan), Hematopoietic Stem Cell Transplantation and radiation therapy (Total body Irradiation) mycophenylate mofetil and cyclosporine A.
  Interventions: Drug: Clofarabine; Procedure: Total body Irradiation; Drug: Melphalan; Biological: Hematopoietic Stem Cell Transplantation; Drug: Alemtuzumab; Drug: mycophenylate mofetil; Device: Cyclosporine A; Drug: Hydroxyurea

INTERVENTIONS:
Drug: Clofarabine — days -7 through -3: 40 mg/m^2 intravenously over 2 hours
  Other Names: Clolar
Procedure: Total body Irradiation — Administration of TBI: The dose of TBI will be 200 cGy given in a single fraction on day -1. The dose rate will be between 10-19 cGy/minute prescribed to the midplane of the patient at the level of the umbilicus.
  Other Names: TLI
Drug: Melphalan — day -2: 140 mg/m^2 intravenously over 30 minutes
  Other Names: Alkeran
Biological: Hematopoietic Stem Cell Transplantation — receives infusion of stem cells on day 0
Drug: Alemtuzumab — 0.3 mg/kg intravenously (IV) days -12 through -8
  Other Names: Campath 1-H
Drug: mycophenylate mofetil — Day -3 through Day 30: 1 gram three times daily (total daily dose 3 grams/day) if the recipient is >50 kg, or 15 mg/kg three times daily if the recipient is ≤50 kg. The same dosage is used orally or intravenously. Consider dose modification if renal impairment (GFR<25 mL/minute corrected)
  Other Names: MMF
Device: Cyclosporine A — Patients will receive CsA therapy beginning on day -3. Dosing of CsA will be 2.5 mg/kg/dose intravenously (IV); if the recipient body weight is <40 kg, dosing will be 3 times daily, and if > 40 kg twice daily. An attempt will be made to maintain a trough cyclosporine level of 250 mg/L to 350 mg/L. Once the patient can tolerate oral medications and has a normal gastrointestinal transit time, CsA will be converted to an oral form at a dose 2.5 x the current IV dose (maximum 12.5 mg/kg/day as initial oral dose).
  CsA taper begins at day +100.
  Other Names: CsA
Drug: Hydroxyurea — hydroxyurea (HU) beginning day -28 and continuing through alemtuzumab administration
  Other Names: Hydria; HU

SUMMARY:
Hematopoietic stem cell transplantation has proven effective therapy for individuals with adrenoleukodystrophy (ALD), metachromatic leukodystrophy (MLD) or globoid cell leukodystrophy (GLD, or Krabbe disease). This protocol also considers other inherited metabolic diseases such as, but not limited to, GM1 gangliosidosis, Tay Sachs disease, Sanfilippo syndrome or Sandhoff disease, I-cell disease (mucolipidosis II).

For patients with advanced or rapidly progressive disease, the morbidity and mortality with transplantation is unacceptably high. Unfortunately, there are no viable alternative therapeutic options for these patients; if transplantation is not performed the patients are sent home to die. Our group at Minnesota has developed a new protocol incorporating transplantation using a reduced intensity conditioning regimen designed to decrease toxicity associated with the transplant procedure. This regimen will make use of the drug clofarabine, which has lympholytic and immune suppressive properties without the neurologic toxicity observed in the related compound, fludarabine, commonly used for transplantation. In addition, several agents providing anti-oxidant and anti-inflammatory properties will be used to assist in the stabilization of the disease processes. This revised transplant protocol will test the following: 1) the ability to achieve engraftment with the reduced intensity protocol, 2) the mortality associated with transplant by day 100, 3) patient outcomes, based on differential neurologic, neuropsychologic, imaging and biologic evaluations prior to transplantation and at designated points after transplantation (day 100, 6 months, 1, 2 and 5 years). Additional biologic studies will include pharmacokinetics of clofarabine and mycophenolate mofetil (MMF). In addition, for patients undergoing lumbar puncture studies, cerebrospinal fluid (CSF) will be requested for determinations of biologic parameters.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation has proven effective therapy for individuals with adrenoleukodystrophy (ALD), metachromatic leukodystrophy (MLD) or globoid cell leukodystrophy (GLD, or Krabbe disease). However, for patients with advanced or rapidly progressive disease, the morbidity and mortality with transplantation is unacceptably high. Unfortunately, there are no viable alternative therapeutic options for these patients; if transplantation is not performed the patients are sent home to die. Our group at Minnesota has developed a new protocol incorporating transplantation using a reduced intensity conditioning regimen designed to decrease toxicity associated with the transplant procedure. This regimen will make use of the drug clofarabine, which has lympholytic and immune suppressive properties without the neurologic toxicity observed in the related compound, fludarabine, commonly used for transplantation. In addition, several agents providing anti-oxidant and anti-inflammatory properties will be used to assist in the stabilization of the disease processes. This revised transplant protocol will test the following: 1) the ability to achieve engraftment with the reduced intensity protocol, 2) the mortality associated with transplant by day 100, 3) patient outcomes, based on differential neurologic, neuropsychologic, imaging and biologic evaluations prior to transplantation and at designated points after transplantation (day 100, 6 months, 1, 2 and 5 years). Additional biologic studies will include pharmacokinetics of clofarabine and mycophenolate mofetil (MMF), develop experience in kinetics of N-acetylcysteine, and evaluate biologic markers of oxidative status during transplantation. In addition, for patients undergoing lumbar puncture studies, cerebrospinal fluid (CSF) will be requested for determinations of biologic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adrenoleukodystrophy: Patients from 0-55 years of age diagnosed with ALD as determined by very long chain fatty acid testing will be eligible for this protocol if they have evidence of cerebral or cerebellar disease based on MRI testing, AND they are determined high risk for any of the following reasons:

  1. Age >18 years
  2. MRI score >10
  3. Evidence of aggressive disease that in the judgment of the Inherited Metabolic and Storage Disease group is sufficiently concerning to consider transplantation with a reduced intensity regimen instead of a standard full preparative regimen.
* Metachromatic Leukodystrophy: Patients from 0-55 years of age diagnosed with MLD as determined by determinations of arylsulfatase A testing will be eligible for this protocol IF they are determined high risk for any of the following reasons:

  1. Age >18 years
  2. Symptomatic disease, as based on neurologic examination, or evidence of deterioration based on subsequent neuropsychologic evaluations.
  3. Evidence of aggressive disease such as rapidly changing MRI determinations that in the judgment of the Inherited Metabolic and Storage Disease group is sufficiently concerning to consider transplantation with a reduced intensity regimen instead of a standard full preparative regimen.
* Globoid Cell Leukodystrophy: Patients from 0-55 years of age diagnosed with GLD as determined by determinations of galactocerebrosidase testing will be eligible for this protocol IF they are determined high risk for any of the following reasons:

  1. Age >18 years
  2. Symptomatic disease, as based on neurologic examination, or evidence of deterioration based on subsequent neuropsychologic evaluations.
  3. Evidence of aggressive disease such as rapidly changing MRI determinations that in the judgment of the Inherited Metabolic and Storage Disease group is sufficiently concerning to consider transplantation with a reduced intensity regimen instead of a standard full preparative regimen.
* Patients with GM1 gangliosidosis, Tay Sachs disease, Sanfilippo syndrome, Wolman disease or Sandhoff disease or other inherited metabolic diseases including but not limited to I-cell disease (mucolipidosis II) who are determined to be sufficiently advanced or high risk based on the following reasons:

  1. Symptomatic disease, as based on neurologic examination, or evidence of deterioration based on subsequent neuropsychologic evaluations.
  2. Evidence of an expected poor outcome based on genetic testing or a prior family history of aggressive disease.
  3. Other metabolic disorders, including but not limited to I-cell disease, that are deemed to be high-risk for a poor outcome with a standard transplant regimen due to anticipated toxicity based on experience gained at the University of Minnesota or other centers.

Exclusion criteria:

* Major organ dysfunction.
* Advanced Disease Exclusion: Following evaluation, if a consensus of the members of the Inherited Metabolic and Storage Disease Program is that a patient is too advanced to benefit in a measurable and meaningful way from transplant, this will be communicated to the family, and transplant will not be offered. Measures to assist in those determinations may include: neurologic/neurocognitive functions such as activities of daily living, motor function, vision, hearing, interaction with environment, toileting, swallowing, or other standardized measures

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Miller WP, Rothman SM, Nascene D, Kivisto T, DeFor TE, Ziegler RS, Eisengart J, Leiser K, Raymond G, Lund TC, Tolar J, Orchard PJ. Outcomes after allogeneic hematopoietic cell transplantation for childhood cerebral adrenoleukodystrophy: the largest single-institution cohort report. Blood. 2011 Aug 18;118(7):1971-8. doi: 10.1182/blood-2011-01-329235. Epub 2011 May 17. PMID 21586746

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Patients: Patients receiving chemotherapy (Hydroxyurea, Alemtuzumab, Clofarabine, Melphalan), Hematopoietic Stem Cell Transplantation and radiation therapy (Total body Irradiation) mycophenylate mofetil and cyclosporine A.
  Clofarabine: days -7 through -3: 40 mg/m^2 intravenously over 2 hours
  Total body Irradiation: Administration of TBI: The dose of TBI will be 200 cGy given in a single fraction on day -1. The dose rate will be between 10-19 cGy/minute prescribed to the midplane of the patient at the level of the umbilicus.
  Melphalan: day -2: 140 mg/m^2 intravenously over 30 minutes
  Hematopoietic Stem Cell Transplantation: receives infusion of stem cells on day 0
  Alemtuzumab: 0.3 mg/kg intravenously (IV) days -12 through -8
  mycophenylate mofetil: Day -3 through Day 30: 1 gram three times daily (total daily dose 3 grams/day) if the recipient is >50 kg, or 15 mg/kg three times daily if the recipient is ≤50 kg. The same dosage is used orally or intravenously.
Period: Overall Study
Arm/Group | Treated Patients
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treated Patients
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Donor Cell Engraftment
Description: Donor Cell Engraftment is defined as the process of transplanted stem cells reproducing new cells.
Time Frame: Day 100
Population: One patient was not evaluable due to an early death.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 37
Participants | 26

2. Secondary Outcome: Number of Patients Whose Death Was Related to the Transplant
Description: In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 38
Participants | 2

3. Secondary Outcome: Concentrations of Mycophenylate Mofetil (MMF)
Description: MMF levels are to be sent on day +3 to the main laboratory for determinations of MMF kinetics.
  Data was not collected on this outcome measure and is not available for reporting.
Time Frame: Day 3
Population: Data was not collected on this outcome measure and is not available for reporting.
Arm/Group | Treated Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Patients With Acute Graft Versus Host Disease (GVHD)
Description: Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host. Acute GVHD can occur once the donor's cells have engrafted in the transplant recipient. The symptoms typically appear within weeks after transplant.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 38
Participants | 3

5. Secondary Outcome: Number of Patients With Chronic Graft Versus Host Disease (GVHD)
Description: Graft-Versus-Host Disease is a severe complication created by infusion of donor cells into a foreign host. Chronic GVHD can appear at any time after allogeneic transplant or several years after transplant.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 38
Participants | 2

ADVERSE EVENTS:
Arm/Group | Treated Patients
Serious Adverse Events (participants affected / at risk) | 10/38
Other Adverse Events (participants affected / at risk) | 33/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Patients (N=38)
Death Due to Disease Progression (General disorders) | 2
Disease Progression (General disorders) | 4
Infection with Grade 3 or 4 Neutrophils (Infections and infestations) | 1
Graft Failure (General disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Patients (N=38)
Bacterial Infection, Feces (Infections and infestations) | 10
Bacterial Infection, Blood (Infections and infestations) | 12
Pneumonia (Infections and infestations) | 14
Fungal Infection, Skin (Infections and infestations) | 2
Aseptic/Avascular Necrosis, NOS (General disorders) | 2
Bloody Stool (Gastrointestinal disorders) | 2
Capillary Leak (Vascular disorders) | 2
Cerebral and Cerebellar Atrophy (Nervous system disorders) | 2
Requires Hemodialysis, NOS (General disorders) | 2
Hemolytic Anemia (Blood and lymphatic system disorders) | 2
Neuropathy (Nervous system disorders) | 2
Otitis Media (Infections and infestations) | 2
Pneumatosis Coli (Gastrointestinal disorders) | 2
Pulmonary Consolidation (Reproductive system and breast disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Veno-Oclusive Disease (Hepatobiliary disorders) | 2
Fungal Infection, Respiratory (Infections and infestations) | 3
Viral Infection, Skin (Infections and infestations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Requires Myringotomy, NOS (Ear and labyrinth disorders) | 3
Pulmonary Opacities (Respiratory, thoracic and mediastinal disorders) | 3
Sinusitis (Infections and infestations) | 3
Upper Respiratory Infection (Infections and infestations) | 3
Bacterial Infection, Skin (Infections and infestations) | 4
Fungal Infection, Blood (Infections and infestations) | 4
Viral Infection, Feces (Infections and infestations) | 4
Bacterial Infection, Urine (Infections and infestations) | 5
Cystitis, NOS (Renal and urinary disorders) | 5
Viral Infection, Respiratory (Infections and infestations) | 6
Hypertension (Vascular disorders) | 6
Viral Infection, Blood (Infections and infestations) | 7
Pericardial Effusion (Cardiac disorders) | 7
Seizures (Nervous system disorders) | 8
Requires Intubation, NOS (Respiratory, thoracic and mediastinal disorders) | 9

LIMITATIONS AND CAVEATS:
Because the diseases being treated on this study are rare, our intent was to only report these outcomes in context with other protocols.

The data was collected, but is not interpretable without combining the data with additional studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No